CLINICAL TRIAL: NCT05335330
Title: Investigation of Trimester-Specific Normative Values of Biomechanical and Viscoelastic Properties of Thoracolumbar Fascia in Pregnant Women-Pilot Study
Brief Title: Biomechanical and Viscoelastic Properties of Thoracolumbar Fascia in Pregnant Women-Pilot Study
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 34 09/03/2022
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnant Women; First Pregnancy
Keywords: pregnant women; thoracolumbar fascia; stiffness; creep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- First trimester pregnant women (first pregnancy): Pregnant women who are in their first pregnancy and in their first trimester will be evaluated.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Thoracolumbar fascia
- Second trimester pregnant women (first pregnancy): Pregnant women who are in their first pregnancy and in their second trimester will be evaluated.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Thoracolumbar fascia
- Third trimester pregnant women (first pregnancy): Pregnant women who are in their first pregnancy and in their third trimester will be evaluated.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Thoracolumbar fascia

INTERVENTIONS:
Other: Evaluation of biomechanics and viscoelastic properties of Thoracolumbar fascia — The biomechanical and viscoelastic properties of the Thoracolumbar fascia will be measured in the side line position. Measurements will be taken from three different points; L1, L3-4 and L5 level.

SUMMARY:
Pregnancy causes the development of biomechanical adaptations in the musculoskeletal system, especially in the lumbopelvic region. In this context, the thoracolumbar fascia (TLF) is the most important structure in this region and is an exoskeleton for the muscles of the lumbar region. However, it has not been objectively clarified how the TLF adapts to the changes in the lumbopelvic region during pregnancy. Therefore, the aim of this pilot study is to investigate the trimester-specific biomechanical (stiffness, decrement and tone) and viscoelastic (creep and relaxation time) properties of the TLF, which adapts to the lumbopelvic region changes in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* First pregnancy
* They are between the ages of 18-40
* Pre-pregnancy Body-Mass-Index (BMI) < 30 kg/m2

Exclusion Criteria:

* Presence of connective tissue disease
* Deterioration of skin integrity in measurement areas
* Presence of orthopedic, neurological, rheumatic problems that may cause musculoskeletal disorders and deviations from normal in biomechanical alignment
* History of spine, pelvis or lower extremity surgery or fracture in the past 6 months
* Description of chronic (more than 3 months) lumbar-pelvic region pain before pregnancy
* Defining metabolic disorders such as type I, II diabetes, gestational diabetes mellitus (GDM), preeclampsia
* Having Pelvic Girdle Pain

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women at the first pregnancy
Study Population: Pregnant women (first pregnancy)
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the baseline stiffness values of Thoracolumbar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the stiffness (N/m) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side line position.
Evaluation of viscoelastic properties of thoracolumbar fascia | Measurement the baseline relaxation time values of Thoracolumbar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the relaxation time (ms) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side line position.
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the baseline tone values of Thoracolumbar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the tone (Hz) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side line position.
Evaluation of viscoelastic properties of thoracolumbar fascia | Measurement the baseline creep values of Thoracolumb Measurement the baseline creep values of Thoracolumbar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the creep of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side line position.
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the baseline decrement values of Thoracolumbar fascia between 10-14 weeks, between 20-24 weeks and between 32-36 weeks
  Measuring of the decrement of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the side line position.

SECONDARY OUTCOMES:
Evaluation of Body Weight | Measurement the baseline body weight (kg) at evaluation time
  Measuring of the Body Weight
Evaluation of Body Mass Index (BMI) | Measurement the baseline BMI values at evaluation time
  BMI (kg/m2) will be calculated as person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lohr C, Braumann KM, Reer R, Schroeder J, Schmidt T. Reliability of tensiomyography and myotonometry in detecting mechanical and contractile characteristics of the lumbar erector spinae in healthy volunteers. Eur J Appl Physiol. 2018 Jul;118(7):1349-1359. doi: 10.1007/s00421-018-3867-2. Epub 2018 Apr 20. PMID 29679246
- [Background] Hu X, Lei D, Li L, Leng Y, Yu Q, Wei X, Lo WLA. Quantifying paraspinal muscle tone and stiffness in young adults with chronic low back pain: a reliability study. Sci Rep. 2018 Sep 25;8(1):14343. doi: 10.1038/s41598-018-32418-x. PMID 30254233
- [Background] Tincello DG, Teare J, Fraser WD. Second trimester concentration of relaxin and pregnancy related incontinence. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):237-8. doi: 10.1016/s0301-2115(02)00360-3. No abstract available. PMID 12551802
- [Background] Wu Z, Wang Y, Ye Z, Guan Y, Ye X, Chen Z, Li C, Chen G, Zhu Y, Du J, Chen G, Liu W, Xu X. Effects of Age and Sex on Properties of Lumbar Erector Spinae in Healthy People: Preliminary Results From a Pilot Study. Front Physiol. 2021 Sep 20;12:718068. doi: 10.3389/fphys.2021.718068. eCollection 2021. PMID 34616306
- [Background] Sanjana F, Chaudhry H, Findley T. Effect of MELT method on thoracolumbar connective tissue: The full study. J Bodyw Mov Ther. 2017 Jan;21(1):179-185. doi: 10.1016/j.jbmt.2016.05.010. Epub 2016 Jun 3. PMID 28167175